## POSTOPERATIVE GLYCAEMIC CONTROL AND THE SURGICAL SITE INFECTION

## INCIDENCE AMONG LIVER TRANSPLANTATION RECIPIENTS: RANDOMIZED CLINICAL TRIAL

Date: March 13th 2018.

Version: 1

Author:

## Ramon Antonio Oliveira,

Sao Paulo Registered Nurses Board: Number 265.476 RN, MSc, PhD Candidate at University of São Paulo School of Nursing. Graduate Program in Adult Health Nursing.

419, Dr. Eneias de Carvalho Aguiar, Av. Cerqueira César - São Paulo - SP, Brazil.

E-mail: <u>ramon.oliveira@usp.br</u> Phone: +5511987001434

## STATISTICAL ANALYSES PLAN

A Microsoft Excel for Mac 2011® database will be constructed. The data will be typed into two different files to ensure accuracy by an automated check. Afterwards, the data will be transferred to the software Statistical Package for the Social Sciences® for Windows® version 22.0.

The results will be computed with a statistician support, following the research objectives and methods. The following tests will be employed:

- Central tendency and dispersion measures.
- The categorical variables will be analysed by the Pearson's  $\chi^2$  test or Fisher's exact test.
- The continuous variables will be analysed by the Student t-test or Mann-Whitney.
- Survival analysis by Kaplan-Meier estimate and Log-rank test.
- Visual inspection of residuals from QQ plot will be used to determine the normality.
- The significant level adopted will be  $\alpha$ =0,05.